CLINICAL TRIAL: NCT06679413
Title: A Phase 1, Single-Center, Repeat-Dose, Open-Label, Fixed-Sequence Drug-Drug Interaction Study of ZX008 in Healthy Male Or Female Study Participants 18 To 55 Years Of Age
Brief Title: A Study to Assess Drug-drug Interaction of ZX008 in Healthy Male and Female Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP0132
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Healthy Study Participants
Keywords: Healthy Study Participants; fenfluramine HCl; Drug-drug interaction; Phase 1; ZX008
MeSH Terms: interventions — Midazolam; Metformin; Bupropion; Fenfluramine

STUDY DESIGN:
Intervention Model Description: In this single arm study the participants will receive a single dose of the cocktail of probe drugs at the first pre-specified timepoint followed by a washout and repeated oral doses of ZX008 and a single dose of the cocktail of probe drugs at the second pre-specified time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Study participants will receive a single dose of the cocktail of probe drugs at pre-specified timepoints followed by a wash out period. The same study participants will then receive repeated oral doses of fenfluramine HCl (ZX008) and a single dose of the cocktail of probe drugs at pre-specified time points during this Treatment Period.
  Interventions: Drug: midazolam; Drug: metformin; Drug: bupropion; Drug: fenfluramine HCl

INTERVENTIONS:
Drug: midazolam — Study participants will receive a pre specified single oral dose of probe drug midazolam on Day 1 and Day 22 of the study
Drug: metformin — Study participants will receive a pre-specified single oral dose of probe drug metformin on Day 1 and Day 22 of the study
Drug: bupropion — Study participants will receive a pre-specified single oral dose of probe drug bupropion on Day 1 and Day 22 of the study
Drug: fenfluramine HCl — Study participants will receive pre-specified repeated oral doses of fenfluramine HCl (ZX008) from Day 6 to 26 during the study
  Other Names: Fintepla; ZX0008

SUMMARY:
The purpose of the study is to assess the single-dose pharmacokinetics (PK) of 3 probe drugs (midazolam, bupropion, and metformin) before and after repeat doses of ZX008

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive at the time of signing the informed consent form (ICF)
* Body weight of at least 50 kg and body mass index within the range 18 to 32 kg/m^2 (inclusive)
* Male or female
* Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) above 1.1x upper limit of normal (ULN)
* Bilirubin >ULN (isolated bilirubin <1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Participant has clinically significant current or past history of cardiovascular or cerebrovascular disease, such as valvular heart disease, and/or pulmonary hypertension. Participants with any history of stroke or myocardial infarction are excluded.
* Clinically significant history or presence of electrocardiogram (ECG) or echocardiogram (ECHO) findings as judged by the investigator or designee at the Screening Visit and Check-in, including each criterion listed below:
* Abnormal sinus rhythm (heart rate outside of 40bpm and 100bpm)
* QTcF (QT interval corrected using Fridericia's formula) interval >450 msec for male participants or >470 msec for female participants (QTcF is the QT interval corrected for heart rate according to Fridericia's formula, it can be either machine read or manually overread)
* QRS interval >120 msec, confirmed by manual over read
* PR interval >220 msec
* Greater than trace aortic valve regurgitation
* Greater than trace mitral valve regurgitation
* Possible signs of pulmonary arterial hypertension (PAH) with abnormal pulmonary artery systolic pressure (PASP) or PASP >35 mmHg
* Evidence of left ventricular dysfunction (systolic or diastolic)
* Clinically significant structural cardiac abnormality, including, but not limited to, mitral valve prolapse, atrial or ventricular septal defects, and patent ductus arteriosus with reversal of shunt (right to left shunt). Note: Patent foramen ovale or a bicuspid aortic valve is not considered exclusionary
* Clinically significant abnormal blood pressure (as determined by the investigator)
* Participant has a current or past history of glaucoma
* Participant has used hepatic enzyme-inducing drugs (eg, glucocorticoids, phenobarbital, isoniazid, phenytoin, rifampicin) within 30 days before the first administration of the cocktail of 3 probe drugs (metformin, midazolam, bupropion) and through the day of discharge from the site
* Participant has used other prescription drugs, including vaccinations, over-the-counter medications, herbal/traditional medicines, or dietary supplements within 14 days before the first administration of the cocktail of probe drugs (excluding medicines for external use), with the exception of acetaminophen (up to 2 g/day)
* Consent to genotyping is required for participation in the study. Poor metabolizers of CYP (cytochrome P450) 3A4 or CYP2B6 based on genotyping and as categorized by the testing laboratory will be excluded from the study
* Positive test for alcohol and/or prohibited concomitant drugs (including cotinine) at Screening Visit and on Day -1
* Participant has donated blood or plasma or has experienced blood loss ≥500 mL within 90 days, ≥200 mL within 30 days, or has donated any blood or plasma within 14 days before first administration of study treatments
* Any consumption of food products with a known Drug-drug interaction (DDI) impact (eg, grapefruit, grapefruit juice, Seville oranges, or products containing them) for at least 1 week before Day 1 and through day of discharge from the site
* Consumption of more than 600 mg of caffeine/day (1 cup of coffee contains approximately 100 mg of caffeine, 1 cup of tea approximately 30 mg, and 1 glass of cola approximately 20 mg) within 30 days before Day 1 and through day of discharge from the site
* Participant is a current smoker or has used nicotine-containing products (eg, tobacco, patches, gum, vapes, or e-cigarettes) within 35 days before Day 1 and through day of discharge from the site

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of midazolam administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple specified time points (up to 96 hours) postdose
  Cmax=Maximum concentration.
Maximum concentration (Cmax) of metformin administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple specified time points (up to 96 hours) postdose
  Cmax=Maximum concentration.
Maximum concentration (Cmax) of bupropion administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple specified time points (up to 96 hours) postdose
  Cmax=Maximum concentration.
Area under the curve from 0 to infinity (AUC) of midazolam administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple time points (up to 96 hours) postdose
  AUC=Area under the curve from 0 to infinity.
Area under the curve from 0 to infinity (AUC) of metformin administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple time points (up to 96 hours) postdose
  AUC=Area under the curve from 0 to infinity.
Area under the curve from 0 to infinity (AUC) of bupropion administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple time points (up to 96 hours) postdose
  AUC=Area under the curve from 0 to infinity.
Area under the curve from 0 to the time of the last quantifiable concentration AUC(0-t) of midazolam administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple time points (up to 96 hours) postdose
  AUC(0-t)=Area under the curve from 0 to the time of the last quantifiable concentration.
Area under the curve from 0 to the time of the last quantifiable concentration AUC(0-t) of metformin administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple time points (up to 96 hours) postdose
  AUC(0-t)=Area under the curve from 0 to the time of the last quantifiable concentration.
Area under the curve from 0 to the time of the last quantifiable concentration AUC(0-t) of bupropion administered alone | Plasma samples will be collected starting from Day 1 at predose and at multiple time points (up to 96 hours) postdose
  AUC(0-t)=Area under the curve from 0 to the time of the last quantifiable concentration.
Maximum concentration (Cmax) of midazolam after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple specified time points (up to 96 hours) postdose of midazolam
  Cmax=Maximum concentration.
Maximum concentration (Cmax) of metformin after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple specified time points (up to 96 hours) postdose of metformin
  Cmax=Maximum concentration.
Maximum concentration (Cmax) of bupropion after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple specified time points (up to 96 hours) postdose of bupropion
  Cmax=Maximum concentration.
Area under the curve from 0 to infinity (AUC) of midazolam after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple time points (up to 96 hours) postdose of midazolam
  AUC=Area under the curve from 0 to infinity.
Area under the curve from 0 to infinity (AUC) of metformin after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple time points (up to 96 hours) postdose of metformin
  AUC=Area under the curve from 0 to infinity.
Area under the curve from 0 to infinity (AUC) of bupropion after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple time points (up to 96 hours) postdose of bupropion
  AUC=Area under the curve from 0 to infinity.
Area under the curve from 0 to the time of the last quantifiable concentration AUC(0-t) of the cocktail of midazolam after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple time points (up to 96 hours) postdose of midazolam
  AUC(0-t)=Area under the curve from 0 to the time of the last quantifiable concentration.
Area under the curve from 0 to the time of the last quantifiable concentration AUC(0-t) of metformin after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple time points (up to 96 hours) postdose of metformin
  AUC(0-t)=Area under the curve from 0 to the time of the last quantifiable concentration.
Area under the curve from 0 to the time of the last quantifiable concentration AUC(0-t) of bupropion after ZX008 administration | Plasma samples will be collected starting from Day 22 at predose and at multiple time points (up to 96 hours) postdose of bupropion
  AUC(0-t)=Area under the curve from 0 to the time of the last quantifiable concentration.

SECONDARY OUTCOMES:
Percentage of study participants with treatment-emergent adverse events (TEAEs) | From Baseline (Day 1) to the end of Safety Follow-Up (up to 116 days)
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0132 1001, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.